CLINICAL TRIAL: NCT00643994
Title: Prospective Evaluation of CyberKnife Stereotactic Radiosurgery for Low and Intermediate Risk Prostate Cancer: Homogenous Dose Distribution
Brief Title: CyberKnife Radiosurgery for Organ-Confined Prostate Cancer: Homogenous Dose Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accuray Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCP001.4
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Prostatic Cancer; Prostate Neoplasms; Prostatic Neoplasms; Cancer of the Prostate
Keywords: Prostate Cancer; CyberKnife; Stereotactic Radiosurgery; Radiotherapy; Radiation; Prostate Tumor; Prostate Surgery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyberKnife Stereotactic Radiosurgery (Experimental): 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction in patients with low and intermediate risk prostate cancer.
  Interventions: Radiation: CyberKnife Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Radiosurgery — 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction
  Other Names: CyberKnife

SUMMARY:
The purpose of this study is to determine the effects of CyberKnife radiosurgery in patients with early stage organ-confined prostate cancer.

DETAILED DESCRIPTION:
The CyberKnife Robotic Radiosurgery System is a unique radiosurgical system capable of treating tumors anywhere in the body noninvasively and with sub-millimeter accuracy. The CyberKnife System delivers radiation using a precise targeting methodology allowing a focal treatment margin around the target, thus limiting the volume of adjacent tissue receiving high doses radiation. This in turn allows the delivery of high doses of radiation to the prostate over a short series of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Histologically proven prostate adenocarcinoma
* Patients belonging in one of the following risk groups:

Low: Clinical Stage (CS) T1b-T2a and Gleason 2-6 and Prostate Specific Antigen (PSA) ≤ 10, or Intermediate: CS T2b and Gleason 2-6 and PSA ≤ 10 or CS T1b-T2b, and Gleason 2-6 and PSA ≤ 20 ng/ml or Gleason 7 and PSA ≤ 10 ng/ml

* Prostate volume: ≤ 100 cc
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Prior prostatectomy or cryotherapy of the prostate
* Prior radiotherapy to the prostate or lower pelvis
* Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion
* Chemotherapy for a malignancy in the last 5 years
* History of an invasive malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years.
* Hormone ablation for two months prior to enrollment, or during treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2007-12; Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Meier, MD, Study Chair — Swedish Cancer Center; Irving Kaplan, MD, Study Chair — Beth Israel Deaconess Medical Center; Martin Sanda, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (23):
- United States (23):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Scripps Cancer Center - CyberKnife of Southern California at Vista, La Jolla, California
  - The CyberKnife at Newport Diagnostic Center, Newport Beach, California
  - Georgetown University, Washington D.C., District of Columbia
  - Coastal CyberKnife and Radiation Oncology, Ft. Pierce, Florida
  - Jupiter Medical Center & CyberKnife Center of Palm Beach, Jupiter, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Community Cancer Center, Normal, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Lake Saint Louis Oncology, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - St. Mary's Regional Medical Center, Reno, Nevada
  - Capital Health, Trenton, New Jersey
  - Hematology Oncology Associates of Central New York, Syracuse, New York
  - Virginia Hospital Center, Arlington, Virginia
  - Swedish Cancer Center, Seattle, Washington
  - Southwest Washington Medical Center, Vancouver, Washington
  - Southwest Washington Regional Cancer Center, Vancouver, Washington
  - ThedaCare Appleton Medical Center, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meier RM, Bloch DA, Cotrutz C, Beckman AC, Henning GT, Woodhouse SA, Williamson SK, Mohideen N, Dombrowski JJ, Hong RL, Brachman DG, Linson PW, Kaplan ID. Multicenter Trial of Stereotactic Body Radiation Therapy for Low- and Intermediate-Risk Prostate Cancer: Survival and Toxicity Endpoints. Int J Radiat Oncol Biol Phys. 2018 Oct 1;102(2):296-303. doi: 10.1016/j.ijrobp.2018.05.040. Epub 2018 Jun 1. PMID 30191864
- See also: Accuray Website — http://www.accuray.com

RESULTS

PARTICIPANT FLOW:
Groups:
- CyberKnife Stereotactic Radiosurgery: Low and intermediate risk patients received 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction
Period: Overall Study
Arm/Group | CyberKnife Stereotactic Radiosurgery
Started (Received CyberKnife 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction) | 310 (379 patients signed the informed consent form and were enrolled. Of these 379 patients, 69 did not participate in the study due to not meeting eligibility criteria, insurance did not approve participation in a clinical study, or the patient withdrew from study prior to receiving treatment.)
10-yr Follow up (optional extension per protocol amendment) | 69
Completed (Completed required 5-year follow up) | 214
Not Completed | 96
Not completed — Death | 24
Not completed — Lost to Follow-up | 72

BASELINE CHARACTERISTICS:
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 310
Age, Continuous [Mean (Full Range); unit: years] — Age at time of CK treatment
  years | 67.6 [41.1 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 310
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Black/African American | 18
  Hispanic/Latino | 5
  Native Hawaiian or Other Pacific Islander | 1
  White | 280
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 310
Clinical Stage (Tumor) [Count of Participants; unit: Participants] — Clinical T category of prostate cancer, estimated by investigator at the time of patient screening.
  Participants
    T1b = Tumor incidental histological finding in >5% of tissue resected | 3
    T1c = Tumor identified by needle biopsy found in one or both sides, but not palpable | 244
    T2a = Tumor involves ½ of one side or less | 54
    T2b = Tumor involves >½ of one side but not both sides | 9
Total Gleason Score [Count of Participants; unit: Participants] — The Gleason score is calculated by adding together the two grades of cancer cells that make up the largest areas of the biopsied tissue sample. The Gleason score usually ranges from 6 to 10. Cancer cells that look similar to healthy cells receive a low score. Cancer cells that look less like healthy cells or look more aggressive receive a higher score.
  Patients with Gleason scores 2-6 are in the Low Risk Group. Patients with Gleason scores of 7 are in the Intermediate Risk Group.
  Participants
    Gleason 2 - 6 | 181
    Gleason 7 | 129
Prostate Specific Antigen (PSA) [Mean (Full Range); unit: ng/mL] | 5.53 [0.04 to 17.90]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  It was developed by the ECOG and published in 1982.
  Participants
    0 = Fully active, able to carry on all pre-disease performance without restriction | 293
    1 = Restricted in physically strenuous activity | 10
    2 = Capable of all selfcare but unable to carry out any work activities | 0
    3 = Capable of only limited selfcare | 1
    Unreported | 6
American Joint Committee on Cancer (AJCC) 6th Edition Risk Group [Count of Participants; unit: Participants]
  Low: Clinical Stage (CS) T1b-T2a, Gleason 2-6, Prostate Specific Antigen (PSA) ≤ 10 ng/ml | 172
  Intermediate: CS T2b, Gleason 2-6, PSA ≤ 10 ng/ml | 1
  Intermediate: CS T1b-T2b, and Gleason 2-6, PSA ≤ 20 ng/ml | 37
  Intermediate: CS T1b-T2b and Gleason 7, PSA ≤ 10 ng/ml | 100

OUTCOME MEASURES:

1. Primary Outcome: Risk for Gastrointestinal (GI) and Genitourinary (GU) Toxicity
Description: To estimate the rates of acute and late Grade 3-5 gastrointestinal and genitourinary toxicities (adverse events [AE]) observed during the 5 years following CyberKnife (CK) treatment for prostate cancer. Kaplan Meier estimates for 5-yr and 10-yr are reported.
  Adverse events occurring within 3 months of treatment were categorized as acute toxicities, and those developing after 3 months were considered late toxicities.
  The rates were determined using the first Grade 3 or higher adverse event per patient, reported as possibly, probably, or definitely related to CK treatment.
  The Common Toxicity Criteria for Adverse Events (CTCAE) Version 3.0 was used to determine the Grade or severity of adverse events in this study, with Grade 3 being severe or medically significant but not immediately life-threatening, Grade 4 being life-threatening and Grade 5 being death related to the adverse event.
Time Frame: Primary Safety Endpoint was measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 310
percentage of participants
  Probability of experiencing Acute GI Grade 3+ event(s) | 0
  Probability of experiencing Acute GU Grade 3+ event(s) | 0
  Probability of experiencing Late GI Grade 3+ events 5 years post treatment | 0
  Probability of experiencing Late GU Grade 3+ events 5 years post treatment | 1.5
  Probability of experiencing Late GI Grade 3+ event(s) at 10 years post CK treatment | 0
  Probability of experiencing Late GU Grade 3+ event(s) at 10 years post CK treatment | 1.5

2. Primary Outcome: Biochemical Disease-Free Survival (bDFS)
Description: To determine the rate of biochemical Disease-Free Survival (bDFS), using the Phoenix definition, following CyberKnife treatment. Kaplan Meier estimates for 5-yr and 10-yr are reported.
  The Phoenix definition uses a Prostate Specific Antigen (PSA) value exceeding the patient's lowest PSA value (nadir) + 2 ng/mL as an indicator of disease recurrence. The percentage of patients who did not have such a PSA rise or receive any interventional therapy to treat prostate cancer are reported below.
Time Frame: Primary Efficacy Endpoint was measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 310
percentage of participants
  Probability of remaining disease-free at 5 years post-CyberKnife treatment | 97.3
  Probability of remaining disease-free at 10 years post-CyberKnife treatment | 91.7

3. Secondary Outcome: Disease Control and Survival Outcomes
Description: To determine the rates of local failure, distant failure, disease-free survival, disease-specific survival, and overall survival following CyberKnife treatment in prostate cancer patients. Kaplan Meier estimates for 5-yr and 10-yr are reported.
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 310
percentage of participants
  Probability of remaining free from Local Failure at 5 years post-CyberKnife treatment | 99.7
  Probability of remaining free from Local Failure at 10 years post-CyberKnife treatment | 96.4
  Probability of remaining free from Distant Failure at 5 years post-CyberKnife treatment | 99.3
  Probability of remaining free from Distant Failure at 10 years post-CyberKnife treatment | 98.6
  Probability of remaining free from disease at 5 years post-CyberKnife treatment | 97.3
  Probability of remaining free from disease at 10 years post-CyberKnife treatment | 90.1
  Probability of remaining free from prostate cancer at 5 years post-CyberKnife treatment | 100
  Probability of remaining free from prostate cancer at 10 years post-CyberKnife treatment | 100
  Probability of Overall survival at 5 years post-CyberKnife treatment | 95.7
  Probability of Overall survival at 10 years post-CyberKnife treatment | 83.8

4. Secondary Outcome: Quality of Life Assessments: American Urological Association (AUA) Symptom Index (SI)
Description: AUA-SI is a 7-item self-report measure used to assess urinary urgency, frequency, and voiding symptoms with scores ranging from 0 (no symptom) to 5 (symptom occurs almost always).
  Total score: 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: AUA questionnaires were completed by patients for milestone follow-up visits, with 306/310 patients completing a baseline questionnaire. All questions needed to be completed in order to calculate the score. Scores obtained per instructions (if possible) and analyzed even if questionnaires were received/dated outside protocol specified visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 306
score on a scale
  Baseline | 7.58 (5.97)
  Last Day of Treatment: number analyzed (Participants) | 297
  Last Day of Treatment | 12.53 (8.11)
  1 Week Post Treatment: number analyzed (Participants) | 300
  1 Week Post Treatment | 14.13 (8.29)
  1 Month Post Treatment: number analyzed (Participants) | 299
  1 Month Post Treatment | 11.64 (7.30)
  3 Months Post Treatment: number analyzed (Participants) | 296
  3 Months Post Treatment | 7.53 (5.54)
  6 Months Post Treatment: number analyzed (Participants) | 292
  6 Months Post Treatment | 7.20 (5.71)
  12 Months Post Treatment: number analyzed (Participants) | 283
  12 Months Post Treatment | 8.49 (6.48)
  18 Months Post Treatment: number analyzed (Participants) | 275
  18 Months Post Treatment | 7.84 (6.27)
  24 Months Post Treatment: number analyzed (Participants) | 271
  24 Months Post Treatment | 7.32 (5.69)
  36 Months Post Treatment: number analyzed (Participants) | 239
  36 Months Post Treatment | 6.59 (5.73)
  48 Months Post Treatment: number analyzed (Participants) | 215
  48 Months Post Treatment | 6.41 (5.90)
  60 Months Post Treatment: number analyzed (Participants) | 200
  60 Months Post Treatment | 6.13 (6.17)
  72 Months Post Treatment: number analyzed (Participants) | 117
  72 Months Post Treatment | 5.62 (5.93)
  84 Months Post Treatment: number analyzed (Participants) | 107
  84 Months Post Treatment | 5.77 (5.85)
  96 Months Post Treatment: number analyzed (Participants) | 94
  96 Months Post Treatment | 4.97 (6.25)
  108 Months Post Treatment: number analyzed (Participants) | 81
  108 Months Post Treatment | 4.60 (5.35)
  120 Months Post Treatment: number analyzed (Participants) | 62
  120 Months Post Treatment | 4.79 (5.33)

5. Secondary Outcome: Quality of Life Assessments: Expanded Prostate Cancer Index Composite (EPIC) -26 Urinary Incontinence
Description: EPIC-26 is a short form version of the Expanded Prostate Cancer Index Composite, and is a validated comprehensive instrument developed to measure the health-related quality of life among men with prostate cancer. EPIC-26 consists of 26 items under 5 domains of urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal.
  Answers qualitatively measure patient's bother for each symptom and are then normalized on a scale of 0 (worst) to 100 (best) to calculate domain scores if sufficient input is provided.
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: EPIC questionnaires were completed by patients at follow-up visits, with 300/310 patients completing a baseline questionnaire. A minimum number of questions needed to be completed within each domain in order to calculate a domain score. Domain scores obtained per instructions (if possible) and analyzed even if questionnaires were received/dated outside protocol specified visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 300
score on a scale
  Baseline | 94.03 (11.69)
  1 Month Post Treatment: number analyzed (Participants) | 296
  1 Month Post Treatment | 89.30 (16.13)
  6 Months Post Treatment: number analyzed (Participants) | 284
  6 Months Post Treatment | 92.08 (14.70)
  12 Months Post Treatment: number analyzed (Participants) | 280
  12 Months Post Treatment | 88.49 (17.16)
  24 Months Post Treatment: number analyzed (Participants) | 267
  24 Months Post Treatment | 89.03 (18.30)
  36 Months Post Treatment: number analyzed (Participants) | 225
  36 Months Post Treatment | 89.23 (18.33)
  48 Months Post Treatment: number analyzed (Participants) | 194
  48 Months Post Treatment | 88.39 (17.85)
  60 Months Post Treatment: number analyzed (Participants) | 173
  60 Months Post Treatment | 89.04 (17.36)
  72 Months Post Treatment: number analyzed (Participants) | 100
  72 Months Post Treatment | 89.84 (19.18)
  84 Months Post Treatment: number analyzed (Participants) | 86
  84 Months Post Treatment | 89.46 (17.42)
  96 Months Post Treatment: number analyzed (Participants) | 71
  96 Months Post Treatment | 90.79 (15.96)
  108 Months Post Treatment: number analyzed (Participants) | 62
  108 Months Post Treatment | 90.28 (17.13)
  120 Months Post Treatment: number analyzed (Participants) | 54
  120 Months Post Treatment | 89.42 (17.15)

6. Secondary Outcome: Quality of Life Assessments: EPIC-26 Urinary Irritative Obstructive
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 300
score on a scale
  Baseline | 87.85 (12.56)
  1 Month Post Treatment: number analyzed (Participants) | 296
  1 Month Post Treatment | 75.20 (18.37)
  6 Months Post Treatment: number analyzed (Participants) | 284
  6 Months Post Treatment | 87.82 (13.76)
  12 Months Post Treatment: number analyzed (Participants) | 280
  12 Months Post Treatment | 84.29 (16.57)
  24 Months Post Treatment: number analyzed (Participants) | 267
  24 Months Post Treatment | 87.43 (13.63)
  36 Months Post Treatment: number analyzed (Participants) | 225
  36 Months Post Treatment | 89.64 (11.85)
  48 Months Post Treatment: number analyzed (Participants) | 194
  48 Months Post Treatment | 88.76 (13.45)
  60 Months Post Treatment: number analyzed (Participants) | 173
  60 Months Post Treatment | 90.36 (12.66)
  72 Months Post Treatment: number analyzed (Participants) | 100
  72 Months Post Treatment | 92.57 (10.41)
  84 Months Post Treatment: number analyzed (Participants) | 86
  84 Months Post Treatment | 92.11 (10.65)
  96 Months Post Treatment: number analyzed (Participants) | 71
  96 Months Post Treatment | 90.77 (12.29)
  108 Months Post Treatment: number analyzed (Participants) | 62
  108 Months Post Treatment | 91.70 (9.78)
  120 Months Post Treatment: number analyzed (Participants) | 54
  120 Months Post Treatment | 92.28 (9.24)

7. Secondary Outcome: Quality of Life Assessments: EPIC-26 Bowel
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 300
score on a scale
  Baseline | 94.88 (9.66)
  1 Month Post Treatment: number analyzed (Participants) | 296
  1 Month Post Treatment | 83.47 (18.83)
  6 Months Post Treatment: number analyzed (Participants) | 284
  6 Months Post Treatment | 91.61 (13.42)
  12 Months Post Treatment: number analyzed (Participants) | 280
  12 Months Post Treatment | 90.12 (14.60)
  24 Months Post Treatment: number analyzed (Participants) | 267
  24 Months Post Treatment | 92.18 (13.00)
  36 Months Post Treatment: number analyzed (Participants) | 225
  36 Months Post Treatment | 92.88 (11.67)
  48 Months Post Treatment: number analyzed (Participants) | 194
  48 Months Post Treatment | 92.52 (12.89)
  60 Months Post Treatment: number analyzed (Participants) | 173
  60 Months Post Treatment | 92.42 (12.63)
  72 Months Post Treatment: number analyzed (Participants) | 100
  72 Months Post Treatment | 94.31 (9.79)
  84 Months Post Treatment: number analyzed (Participants) | 86
  84 Months Post Treatment | 94.29 (10.08)
  96 Months Post Treatment: number analyzed (Participants) | 71
  96 Months Post Treatment | 93.44 (9.46)
  108 Months Post Treatment: number analyzed (Participants) | 62
  108 Months Post Treatment | 92.89 (9.73)
  120 Months Post Treatment: number analyzed (Participants) | 54
  120 Months Post Treatment | 93.77 (8.93)

8. Secondary Outcome: Quality of Life Assessments: EPIC-26 Sexual
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyberKnife Stereotactic Radiosurgery
Number analyzed (Participants) | 300
score on a scale
  Baseline | 56.79 (31.95)
  1 Month Post Treatment: number analyzed (Participants) | 296
  1 Month Post Treatment | 53.74 (31.47)
  6 Months Post Treatment: number analyzed (Participants) | 284
  6 Months Post Treatment | 53.74 (33.49)
  12 Months Post Treatment: number analyzed (Participants) | 280
  12 Months Post Treatment | 50.19 (32.83)
  24 Months Post Treatment: number analyzed (Participants) | 267
  24 Months Post Treatment | 47.71 (32.27)
  36 Months Post Treatment: number analyzed (Participants) | 225
  36 Months Post Treatment | 47.31 (32.36)
  48 Months Post Treatment: number analyzed (Participants) | 194
  48 Months Post Treatment | 46.82 (31.60)
  60 Months Post Treatment: number analyzed (Participants) | 173
  60 Months Post Treatment | 42.88 (31.45)
  72 Months Post Treatment: number analyzed (Participants) | 100
  72 Months Post Treatment | 47.66 (33.93)
  84 Months Post Treatment: number analyzed (Participants) | 86
  84 Months Post Treatment | 48.12 (34.47)
  96 Months Post Treatment: number analyzed (Participants) | 71
  96 Months Post Treatment | 44.16 (30.34)
  108 Months Post Treatment: number analyzed (Participants) | 62
  108 Months Post Treatment | 43.36 (31.36)
  120 Months Post Treatment: number analyzed (Participants) | 54
  120 Months Post Treatment | 50.13 (31.08)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from study enrollment through end of protocol follow-up, including fiducial placement, CyberKnife radiosurgery treatment, and scheduled follow-up visits up to 10 years post-CyberKnife treatment.
Description: All adverse events were collected. Serious Adverse Events reported in clinicaltrials.gov are all events meeting serious criteria regardless of causality.
Arm/Group | CyberKnife Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 21/310
Serious Adverse Events (participants affected / at risk) | 34/310
Other Adverse Events (participants affected / at risk) | 302/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyberKnife Stereotactic Radiosurgery (N=310)
car accident (General disorders) | 1 (1)
Conduction abnormality/ atrioventricular heart block (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Valvular heart disease (Cardiac disorders) | 2 (2)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Death NOS (General disorders) | 9 (9)
Dermatology/skin other - cancer (Skin and subcutaneous tissue disorders) | 2 (2)
GI - other - cancer (Gastrointestinal disorders) | 3 (3)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary/pancreas - other - cancer (Hepatobiliary disorders) | 1 (1)
Hepatobiliary/pancreas - other cirrhosis (Hepatobiliary disorders) | 1 (1)
Infection - heart endocarditis (Infections and infestations) | 1 (1)
infection with unknown ANC (Infections and infestations) | 1 (1)
Potassium serum -low (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal/soft tissue - fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 3 (3)
Neurology - other (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/upper respiratory - cancer (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary obstruction (Renal and urinary disorders) | 1 (1)
Renal/GU - other - cancer (Renal and urinary disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 2 (2)
Other malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
vessel-injury artery - aorta (Vascular disorders) | 1 (1)
GI - other, diverticulosis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyberKnife Stereotactic Radiosurgery (N=310)
Fatigue (General disorders) | 113 (120)
Constipation (Gastrointestinal disorders) | 43 (46)
Diarrhea (Gastrointestinal disorders) | 120 (135)
Flatulence (Gastrointestinal disorders) | 30 (31)
Hemorrhoids (Gastrointestinal disorders) | 16 (17)
Proctitis (Gastrointestinal disorders) | 44 (51)
GI Hemorrhage/Bleeding (Gastrointestinal disorders) | 52 (55) — rectal bleeding, blood in stool
GI Pain (Gastrointestinal disorders) | 25 (25) — Abdominal pain, stomach pain, rectal pain
GU Pain (Renal and urinary disorders) | 184 (231) — Pain with urination (dysuria)
Urinary Incontinence (Renal and urinary disorders) | 28 (38)
Urinary Frequency/Urgency (Renal and urinary disorders) | 232 (332)
Urinary Retention (Renal and urinary disorders) | 157 (190)
Urinary Tract Infection (Renal and urinary disorders) | 14 (15)
GU Hemorrhage/Bleeding (Renal and urinary disorders) | 49 (63) — Blood in urine (hematuria), GU hemorrhage
Back Pain (Musculoskeletal and connective tissue disorders) | 17 (19)
Ejaculatory Dysfunction (Reproductive system and breast disorders) | 16 (17)
Erectile Dysfunction (Reproductive system and breast disorders) | 66 (66)
Sexual/Reproductive Pain (Reproductive system and breast disorders) | 23 (25) — Groin/pelvic pain, pain with ejaculation

LIMITATIONS AND CAVEATS:
A limitation of this study is that of the 21 sites originally enrolling eligible patients, only 14 opted to continue beyond year 5. While 189 patients were followed through year 5, only 135 of these consented to continued follow-up. We also note that several patients were due for their 10-year follow-up during Coronavirus Disease (COVID) lockdowns, hampering study activities such as monitoring visits as well as patient compliance with protocol-required visit windows.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT00643994/Prot_SAP_000.pdf